CLINICAL TRIAL: NCT06287749
Title: French Assessment of Minimal Residual Disease by Liquid Biopsies in Pancreatic Ductal Adenocarcinoma Patients
Brief Title: French Assessment of MRD by Liquid Biopsies in PDAC Patients (FRENCH.MRD.PDAC)
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL23_0298
Record Dates: First submitted 2024-02-08; First posted 2024-03-01 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer Resectable; Pancreatic Ductal Adenocarcinoma; Minimal Residual Disease; Liquid Biopsy; ctDNA
Keywords: Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer Resectable; Minimal Residual Disease; Liquid Biopsy; ctDNA
MeSH Terms: conditions — Neoplasm, Residual | interventions — Blood Specimen Collection; Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ctDNA analysis NGS on tumor specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pancreatic Ductal Adenocarcinoma patients: Resectable PDAC patients
  Interventions: Biological: Blood sample/Liquid Biopsy

INTERVENTIONS:
Biological: Blood sample/Liquid Biopsy — ctDNA analysis

SUMMARY:
The overall objective of this GUIDE.MRD consortium is to confirm that ctDNA detected after curative intended treatment for PDAC is a marker of residual disease and for risk-of-recurrence, and applicable in clinical practice.

Primary objective To confirm that ctDNA analyses performed after PDAC treatment can identify patients with a high risk-of-recurrence.

Specifically, the investigators want to determine the association between disease-free survival (DFS) and ctDNA detection status after

1. curative-intended surgery and
2. adjuvant chemotherapy.

FRENCH.MRD.PDAC is the French study of the european GUIDE.MRD project

DETAILED DESCRIPTION:
PDAC is the most common subtype of pancreatic cancer. The main pillars of non-metastatic PDAC clinical management are (i) surgery and (ii) neoadjuvant treatment including chemotherapy, which can be followed by external radiotherapy in case of borderline/locally advanced tumors.

Adjuvant chemotherapy is standard-of-care and is given to most patients that tolerate it after the extensive surgical procedure. The sequence of perioperative chemotherapy (before, after, both) is currently a matter of debate.

Despite extensive surgical resection and chemotherapy, most patients relapse, and median overall survival in the group of patients that is treated with surgery and modern chemotherapy regimens is below 24 months.

Throughout the body, DNA is released from cells into the circulation. This DNA is collectively referred to as cell-free DNA (cfDNA). In a patient with a solid cancer such as PDAC, a fraction of the cfDNA found in the blood, originates from tumor cells, and is termed circulating tumor DNA (ctDNA).

At present, a multitude of different ctDNA tests are available, and a common standard is lacking. This study is part of the large, EU-funded GUIDE.MRD project that aims to develop international reference standards for ctDNA diagnostics and use the best, standardized tests in clinically meaningful scenarios, including postsurgery follow-up of patients with PDAC, colorectal cancer, and lung cancer.

Detailed Description:

The FRENCH.MRD.PDAC study will prospectively enroll patients in France who undergo potentially curative surgery for PDAC. The intervention is repeated blood sampling at pre-defined time points.

Primary objective To confirm that ctDNA analyses performed after PDAC treatment can identify patients with a high risk-ofrecurrence.

Specifically, the investigators want to determine the association between 3-year disease-free survival (DFS) and ctDNA detection status after

1. curative-intended surgery and
2. adjuvant chemotherapy.

Secondary objectives Secondary objective 1 (S1) To technically assess, compare, and rank existing commercial ctDNA diagnostics after intended curative PDAC treatment (upfront surgery or neoadjuvant treatment followed by surgery +/- postoperative chemotherapy) to identify the best method at each time point, with no impact on diagnosis or treatment of patients enrolled in the study.

Secondary objective 2 (S2) To assess the effect of standard-of-care adjuvant chemotherapy on the level of ctDNA. Especially, for patients with ctDNA detected after surgery, the investigators will measure and compare the ctDNA levels in plasma samples drawn before and after adjuvant chemotherapy. Furthermore, the change in ctDNA level will be correlated to the oncological outcomes (time to clinical recurrence, disease-free survival, and overall survival).

Secondary objective 3 (S3) To investigate if time to Molecular recurrence determined using serial ctDNA analyses in longitudinally collected plasma samples is shorter than time to Clinical recurrence using standard-of-care radiological imaging.

Secondary objective 4 (S4) To investigate the correlation between ctDNA analysis results and findings on CT scans. ctDNA analysis will be restricted to blood sampling times that are coinciding with standard-of-care CT scans. If ctDNA analysis can predict the outcome of the CT scan, the potential is that ctDNA analysis in the future can guide when to perform CT scans.

Secondary objective 5 (S5) To investigate the prognostic power of ctDNA at the time point of indeterminate CT scans.

Patient identification Patients with PDAC are screened for eligibility by the involved physicians based on the protocol of the multidisciplinary tumor board (MDT). The screening will be done based on the electronic health record in the electronic journal (at present, for example, Take Care). The National Health Record may be accessed for some patients to complete the record.

Patient recruitment and informed consent The involved physicians screen patients meeting the inclusion criteria specified below. Eligible patients are approached in person or initially by phone, after they have been informed about the diagnosis and the planned surgery. Patients are given written and oral information about the project by a trained research nurse or by an involved physician. Informed consent will be obtained before the beginning of any study-related procedures.

The signed and dated consent forms are scanned into the project's electronic database and stored physically in a locked space.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic ductal adenocarcinoma, according to the assessment of the MDT.
* Age 18 years or older.
* Scheduled for curative intent surgical resection.

Exclusion Criteria:

* Hereditary pancreatic cancer.
* Verified distant metastases.
* Patients who are unlikely to comply with the protocol (e.g. uncooperative attitude), inability to return for subsequent visits and/or otherwise considered by the Investigator to be unlikely to complete the study.
* Other cancers (excluding prior pancreatic cancer or skin cancer other than melanoma) within 3 years from eligibility screening.
* Pregnant or nursing woman, or in childbearing age and not willing to use contraception
* Adult subject to a legal protection
* Not covered by Health insurance
* Patient unable to understand and sign written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with resected PDAC
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
3-year Disease-free survival (DFS) | 3 years after the end of inclusion
  Disease-free survival was defined as the time between the date of the baseline blood sampling/inclusion and the date of the first event among or recurrence or death from any cause.

SECONDARY OUTCOMES:
Sensitivity (Se) of the ctDNA diagnostics | 3 years after the end of inclusion
  Sensitivity (Se) of the ctDNA diagnostics is calculated in subjects with a 3-year recurrence: Se = TP/(TP+FN) (a positive reference test)
Specificity (Sp) of the ctDNA diagnostics | 3 years after the end of inclusion
  Specificity (Sp) of the ctDNA diagnostics is calculated in subjects without a 3-year recurrence: Sp = TN/(TN+FP) (a negative reference test)
Positive predictive value of the ctDNA diagnostics | 3 years after the end of inclusion
  The predictive value of a positive test or positive predictive value (PPV): PPV = TP/(TP+FP).
Negative predictive value of the ctDNA diagnostics | 3 years after the end of inclusion
  The predictive value of a negative test or negative predictive value (NPV): NPV =TN/(TN+FN).
Are Under the Curve of the ctDNA diagnostics | 3 years atfer the end of inclusion
  Area Under the Curve of the of the ctDNA:
  * AUC ≤0.75 = low classification accuracy,
  * 0.75 < AUC < 0.85 = moderate accuracy,
  * and AUC ≥0.85 = high accuracy
Time to clinical recurrence | 3 years after the end of inclusion
  Time to clinical recurrence was defined as the time between the date of the baseline blood sampling/inclusion [debut] and the date of the recurrence.
Overall survival | 3 years after the end of inclusion
  Overall survival was defined as the time between the date of the baseline blood sampling/inclusion [debut] and the date of death from any cause.
Time to molecular recurrence | 3 years after the end of inclusion
  Time to molecular recurrence was defined as the time between the date of the baseline blood sampling/inclusion [debut] and the date of the molecular recurrence (positive ctDNA test).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas BARDOL, M.D., Principal Investigator — University Hospital, Montpellier; Catherine ALIX-PANABIERES, Ph.D., Study Director — University Hospital, Montpellier
Locations (1):
- CHU de Montpellier, Montpellier, Hérault, France